CLINICAL TRIAL: NCT06604585
Title: The Parental Journey. Digital Tool for Security in Parenthood, a Way to Promote Public Health. A Pilot Study.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 277873
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Primary Prevention; Parenting; Family Relations

STUDY DESIGN:
Intervention Model Description: The pilot study will be conducted as a randomized clinical trial. We will use a two-group design where half of the participants are randomized to the intervention group with access to the digital parent support program and half to the control group with conventional parental support without access to the digital parental support program, 1. Conventional parental support and digital parent support program. (n=15). 2. Conventional parental support (n=15).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention- an interactive digital parental support program in primary care. (Experimental): The intervention group will receive conventional parental support according to the national child health care programme. Additionally, they will have access to the digital parental support program, 'Parenthood - A Journey Together'."
  Interventions: Behavioral: Parenthood - a journey together. Digital tool to increase security in parenthood, a way to promote public health..
- The control group without access to the digital parental support program. (No Intervention): The control group will receive conventional parental support according to the national child health care programme, without access to the digital parental support program, 'Parenthood - A Journey Together'."

INTERVENTIONS:
Behavioral: Parenthood - a journey together. Digital tool to increase security in parenthood, a way to promote public health.. — The project involved the development of an internet-based parental support program to be delivered via the national Support and Treatment (Sob) platform and used in primary care to enhance traditional parental support within child healthcare, as needed. The innovation has been developed in collaboration with the Innovation Fund in Västra Götaland. The aim is to increase the experience of parental competence and a sense of security in parenting by reflecting on attitudes and approaches in interaction with the child through an interactive, digital parental support program. The four themes in the parental support program, "Parenthood a journey together", are named: Being a good enough parent, understanding one's child, interacting with one's child, and meeting daily challenges as a parent regarding food, sleep, play, screen time, and physical activity. The four modules will include explanatory and psychoeducational texts, written exercises, videos, and homework.
  Arms: The intervention- an interactive digital parental support program in primary care.

SUMMARY:
The goal of this randomized clinical pilot study is to evaluate the feasibility and experience of the internet-based parental support program "Parenting - a journey together". This program is intended to be delivered via the national Support and Treatment Platform and used within primary care to enhance traditional parental support within child health care when needed. The main questions it aims to answer are:

1. Is the digital parental support intervention feasible and helpful within primary care?
2. How do parents perceive the program "Parenting - a journey together"?
3. Does the program increase the sense of parental ability and security in parenting by reflecting on attitudes and approaches in interaction with the child?

Participants in this study will be parents of children aged 2-5 years who have expressed interest in participating in the study and in the parental support program. Participants will be randomized into either the intervention group or the control group. Participants will be asked to complete validated questionnaires measuring the parent-child relationship, perceived parental ability, stress, and well-being before and after the parental support program, and again after 3 months. These results will then be compared with those of the control group.The knowledge gained from the pilot study can contribute to the development of digital parental support interventions within primary care. If the pilot study proves that the interactive digital parenting program is feasible for use in child health centers and is perceived as helpful by parents, a larger randomized controlled (RCT) study, (not included in this application) will be conducted to evaluate its effectiveness.

DETAILED DESCRIPTION:
Research question / Hypothesis / Theoretical framework:

Can a digital interactive parental support program be a tool to use within child health care to increase the feeling of security and competence in parenthood?

Additional research questions for the pilot study:

1. What is the percentage of those asked who agree to participate?
2. Can the execution of planned outcome measures be measured practically?
3. Is the intervention practically feasible with the resources that can be expected in a larger study?
4. How many parents terminate their participation in the study after they have been included?
5. How common is the occurrence of unexpected problems?
6. What change is observed between baseline and follow-up measurement of outcome measures in the two different groups?

Study Design:

Quantitative Experimental.

Intervention:

A pilot study will be conducted as a randomized clinical trial to evaluate and investigate whether the digital parent support intervention is feasible within primary care.

Selection Population:

Parents within child health services with children aged 2-5 years. Through a brief presentation of the parent support program and the pilot study in connection with visits to the child health center, where the parents also answer a few short questions, the nurse identifies parents who are interested in participating in the intervention: Parenting - a journey together, digital parent support program.

Method:

Group Division: A two-group design will be used where half are randomized to the intervention group with access to the parent support program and half to the control group with usual parental support without access to the digital parent support program. 1. Usual parental support. (n=15). 2. Usual parental support and digital parent support program. (n=15).

Data Collection:

Parents with children aged 2-5 years within child health services will be recruited to participate in the study. Four child health centers located in different parts of the Västra Götaland region are planned to participate in the recruitment of parents and the different child health centers will also test the intervention. After the parents have accepted participation in the study, all will answer the validated questionnaires that will be used to assess the primary outcome measures. Then a randomization to either intervention group or control group without access to the digital program for comparison is made. Measurement of the primary outcome measures in both groups will also take place after the intervention and 3 months after the intervention. The primary outcome measures include questions about the parent-child relationship, perceived parental capacity, stress and well-being. Surveys planned to be used are: "The Parental Reflective Functioning Questionnaire", "The Parenting Sense of Competence Scale", "The Swedish Parenthood Stress Questionnaire", "The Warwick-Edinburgh Mental Well-being Scale.

Data Processing:

Statistical analysis will be performed to compare the results for the intervention group with the control group. Appropriate statistical tests will be used to evaluate the effect of the digital parental support program on the primary outcome measures from the validated surveys. Descriptive statistics will also be used to present data. In the upcoming main study, the intention is to investigate changes over time in parental experience and the effect of the intervention on this. The same analysis will be performed in the pilot study, although the purpose then is not to demonstrate the effect of the intervention but only to obtain estimates that can facilitate the estimation of the sample size in the upcoming main study. The change in parental experience will be transformed into an ordinal scale with the scale steps improved (+1), unchanged (0), and worsened (-1). If there are few unchanged, the scale steps are transformed into improved (+1) or not improved (0). In the analysis, the transformed change becomes a dependent variable while the participants' gender, participants' age, group affiliation, and follow-up time become fixed independent variables. An interaction variable is also created between group affiliation and follow-up time and this is treated as a fixed effect. The expectation is that a child can have one, two, three, or four parents/partners who undergo the treatment. Randomization takes place per child, and analysis is based on the participants' responses. Each participant is assigned the child's code number. A virtual identification (ID) number will therefore be added for the child as a random effect variable.The statistical analysis becomes a mixed model ordered multivariable logistic regression or mixed model multivariable logistic regression depending on how the investigators choose to treat the dependent variable. The investigators have several outcome measures on parental experience and a separate regression is performed for each outcome measure.

Expected Outcome / Clinical Significance:

By giving parents the opportunity to reflect on their parenting, their interaction with the child, and also practice different ways of handling situations through the individual-based digital program, they are expected to become more confident in their parenting and feel more trust in themselves. This in turn leads to a more favorable environment for the child. The digital parenting support program means increased accessibility to parenting support with a small effort for primary care, and the format makes it possible to scale up to the entire Västra Götaland region. It could also be used nationally as it is on an online platform called "support and treatment". The digital parenting support program is expected to be part of the transformation of primary care for the future.

Project's Gender Perspective:

Traditional parenting support offered in various groups at child health centers and family centers usually attracts mostly mothers and the social profile tends to be more educated parents. This digital program is accessible to both parents and they can work with it when it suits them, which also increases the opportunity to reflect together. Thus, fathers are also involved in a better way than before.

ELIGIBILITY:
Inclusion Criteria:

* Adult parents (or another adult who is a primary caregiver) to children within pediatric healthcare services with children aged 2-5 years old.
* The parents are not participating in other parental support programs or interventions from Child Health Care psychologists, as this would complicate the evaluation of the effects of each intervention.
* Parents who speak Swedish, due to the fact that "Parenting - a journey together" has not yet been translated into other languages.
* Parents who respond affirmatively to the inclusion questions, indicating that they perceive a need for additional parental support and are motivated to participate in the program.

Inclusion questions for assessing a parent's needs and motivation to participate in the digital parenting support program:

1. How important do you consider your ability/confidence as a parent to be for you right now?
2. What has motivated you to consider participating in this program?
3. How motivated are you to make changes in your behavior to improve your parenting ability?
4. Do you have previous experiences with similar digital programs or parental support interventions? If yes, what was your experience?
5. What type of support do you think you need to successfully complete this program?

Exclusion Criteria:

* Parents of children outside the 2-5 years age range. The program is specifically designed for parents within child health care with children in this age group. Once children reach the age of 6, they transition to school health care.
* The parents who are already participating in other parental support programs or receiving interventions from Child Health Care psychologists are not eligible, as this would complicate the evaluation of the effects of each intervention.
* Parents who do not speak Swedish, as the program 'Parenting - a Journey Together' has not yet been translated into other languages.
* Parents who have indicated no perceived need for additional parental support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The Swedish Parenthood Stress Questionnaire - SPSQ | Measurement data is collected at baseline, pre intervention, immediately after the intervention, and 3 months after the intervention.
  The Swedish Parenthood Stress Questionnaire (SPSQ) is designed to measure the perceived stress/strain that parents can directly relate to their parenthood. The questionnaire is influenced by, and primarily originates from parts of R. Abidin's Parenting Stress Index (PSI; Abidin, 1990). In early publications (Östberg, Hagekull, & Wettergren, 1997), SPSQ was referred to as a Swedish PSI (S-PSI) to facilitate comparisons with the American scale. In accordance with an agreement with the American publisher that holds the copyright to the PSI scale, the name has been changed to The Swedish Parenthood Stress Questionnaire (SPSQ). SPSQ is based on 35 selected questions from PSI, with clear and high/acceptable factor loadings (Abidin, 1990). The questions have been selected from the subscales Depression, Restrictions of Role, Sense of Competence, Social Isolation, Relationship with Spouse and Parent Health.
The parental reflective functioning questionnaire- PRFQ | Measurement data is collected at baseline, pre intervention, immediately after the intervention, and 3 months after the intervention.
  The Parental Reflective Functioning Questionnaire (PRFQ) has been developed to provide a brief, multidimensional assessment of parental reflective functioning that is easy to administer to parents with a wide range of socioeconomic and educational backgrounds. Because of the current interest in the role of PRF in the intergenerational transmission of attachment in early childhood, the PRFQ was primarily designed for parents of children 0-5 years of age. The questionnaire consists of 18 items.
The Parenting Sense of Competence scale -PSOC | Measurement data is collected at baseline, pre intervention, immediately after the intervention, and 3 months after the intervention.
  The Parenting Sense of Competence scale (PSOC) is a self-report measure that aims to assesses one's perceived efficacy and satisfaction with parenting. One of the most used scales to measure this construct is Johnston and Mash's version of the Parenting Sense of Competence (PSOC) questionnaire. This scale consists of 16 items and evaluates the caregiver's perceived parenting competence through its two dimensions: efficacy, i.e., the degree to which the parent feels competent in their parenting role and satisfaction, i.e., the extent to which the caregiver feels satisfied with their role as a parent.
Short Warwick Edinburgh Mental Wellbeing Scale -SWEMWBS | Measurement data is collected at baseline, pre intervention, immediately after the intervention, and 3 months after the intervention.
  The Short Warwick Edinburgh Mental Wellbeing scale (SWEMWBS) is a short version of the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS). The WEMWBS was developed to enable the monitoring of mental wellbeing in the general population and the evaluation of projects, programmes and policies which aim to improve mental wellbeing. The SWEMWBS uses seven of the WEMWBS's 14 statements about thoughts and feelings, which relate more to functioning than feelings and so offer a slightly different perspective on mental wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra M Weineland, Ass prof, Study Director — Department of Psychology, Department of medicine, University of Gothenburg .

IPD SHARING:
Plan to Share IPD: Yes
1. Ethical and Legal Considerations:
     Data will be anonymized per data protection laws to safeguard patient privacy. Researchers must sign a data sharing agreement detailing data use, security measures, and confidentiality requirements.
  2. Ethics Committee Approval:
     Documentation of approval from a relevant ethics committee is required to ensure ethical soundness.
  3. Scope and Responsibility:
     Requesters must describe the intended data use and ensure data is not used for other purposes without consent.
     Findings from data use must be shared with us before publication.
  4. Security Measures:
  Researchers must show that appropriate technical and organizational measures are in place for secure data handling and storage.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1. Individual participant data (IPD): Available within 6 months after primary results publication or study completion.
  2. Study Protocol: Available upon request after trial results are published.
  3. Statistical Analysis Plan: Shared upon request post-primary manuscript publication.
  4. Informed Consent Form (ICF): De-identified ICF available upon request post-trial.
  5. Clinical Study Report: Available upon request post-results publication.
  6. Analytic Code:Shared upon request post-primary results publication for transparency.
  Conditions for Access: Formal request and data sharing agreement required. Agreement covers data use, privacy compliance, and ethical standards. Researchers must submit a research plan and ethics approval. PI reviews all requests for compliance.
Access Criteria: 1. Research Proposal: Submit a proposal detailing objectives, methodology, impact, and specific IPD usage.
  2. Ethics Approval: Provide evidence of ethics committee approval confirming ethical soundness.
  3. Data Use Agreement (DUA): Sign a DUA outlining data access terms, including security, confidentiality, and usage limitations.
  4. Data Security Measures: Demonstrate secure IPD handling, including encryption and access controls.
  5. Researcher Qualifications: Provide academic and professional background to ensure research expertise.
  6. Transparency and Accountability: Share results with the data provider before publication and acknowledge the data source.
  7. Purpose Limitation: Use data solely for the specified research purpose.
  8. Publication and Data Sharing: Commit to publishing findings in peer-reviewed journals and sharing results with the scientific community.
  9. Compliance with Regulations: Comply with all applicable data protection laws, including GDPR.

REFERENCES:
- [Background] Luyten P, Mayes LC, Nijssens L, Fonagy P. The parental reflective functioning questionnaire: Development and preliminary validation. PLoS One. 2017 May 4;12(5):e0176218. doi: 10.1371/journal.pone.0176218. eCollection 2017. PMID 28472162
- [Background] Ostberg M, Hagekull B, Wettergren S. A measure of parental stress in mothers with small children: dimensionality, stability and validity. Scand J Psychol. 1997 Sep;38(3):199-208. doi: 10.1111/1467-9450.00028. PMID 9309950
- [Background] Gilmore L, Cuskelly M. Factor structure of the Parenting Sense of Competence scale using a normative sample. Child Care Health Dev. 2009 Jan;35(1):48-55. doi: 10.1111/j.1365-2214.2008.00867.x. Epub 2008 Oct 22. PMID 18991983
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300